CLINICAL TRIAL: NCT04303494
Title: Predictive Value of Heart Rate Variability on Cardiorespiratory Events of Preterm Infants Routinely Immunised in the Hospital
Brief Title: Predictive Value of Heart Rate Variability on Cardiorespiratory Events
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01207; ks17Schulzke
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Post-immunisation Apnoea and Bradycardia of Prematurity (AOP)
MeSH Terms: conditions — Bradycardia | interventions — Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental1: preterm infants will be routinely immunised during primary hospitalisation
  Interventions: Biological: immunisation
- Experimental2: preterm infants discharged and readmitted for immunisation during the 3-year period
  Interventions: Biological: immunisation
- Control: healthy control infants
  Interventions: Biological: immunisation

INTERVENTIONS:
Biological: immunisation — combined diphtheria, tetanus, acellular pertussis, poliomyelitis, hepatitis B, ± Haemophilus influenzae type B and simultaneous pneumococcus (PCV13) vaccination

SUMMARY:
The aim of this study are to investigate whether heart rate variability (HRV) parameters derived from nonlinear time series analysis at five different time points have prognostic utility for assessing the risk of postimmunisation AOP in very preterm/very low birth weight infants immunised in the hospital.

ELIGIBILITY:
Inclusion criteria for preterm infants:

* Gestational Age (GA) 22+0 to 31+6 weeks and/or birth weight 400 g to 1500 g
* Chronological age > 7 days
* Written informed parental consent

Inclusion criteria for term healthy control infants:

* GA 37 to 42 weeks, chronological age 3 to 28 days (beyond initial transition after birth)
* Hospitalised in the neonatal rooming-in unit of the University Children's Hospital Basel as healthy co-twin or healthy sibling, or neonate ready to be discharged home after reconvalescence from minor illness such as hyperbilirubinaemia
* Written informed parental consent

Exclusion Criteria:

* Major congenital malformations including neuromuscular disorders, thoracic malformations, major cardiac malformation
* Lack of written informed parental consent

Ages: 3 Days to 28 Days | Sex: All
Age Groups: Child
Study Population: preterm infants and healthy control infants
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Changes in AOP | record the sum of AOP events from 48 hours windows of raw data, within 24 hours after - 24 hours before immunisation
  Difference in AOP events within 24 hours after - 24 hours before immunisation

SECONDARY OUTCOMES:
Difference in prolonged hypoxaemic episodes | record SpO2 from 48 hours windows of raw data, within 24 hours after - 24 hours before immunisation
  Difference in prolonged hypoxaemic episodes (SpO2 < 80% for at least 1 min) within 24 hours after - 24 hours before immunisation (CAP-trial definition).
Difference in number of manual stimulations | number of manual stimulations within 24 hours after - 24 hours before immunisation
  Difference in number of manual stimulations within 24 hours after - 24 hours before immunisation
Difference in number increases in oxygen concentration | record oxygen concentration from 48 hours windows of raw data, within 24 hours after - 24 hours before immunisation
  Difference in number increases in oxygen concentration within 24 hours after - 24 hours before immunisation
Difference in number of increases in continuous positive airway pressure (CPAP) | within 24 hours after - 24 hours before immunisation
  Difference in number of increases in continuous positive airway pressure (CPAP) within 24 hours after - 24 hours before immunisation
Difference in number of reinstallations in continuous positive airway pressure (CPAP) | within 24 hours after - 24 hours before immunisation
  Difference in number of reinstallations in continuous positive airway pressure (CPAP) within 24 hours after - 24 hours before immunisation
Difference in number of endotracheal intubation | within 24 hours after - 24 hours before immunisation
  Difference in number of endotracheal intubation for AOP events within 24 hours after - 24 hours before immunisation
Difference in sample entropy (SampEn) of interbeat interval of heart rate (IBI) | 24 hours after - immediately prior to immunisation
  Difference in SampEn of IBI 24 hours after - immediately prior to immunisation
Difference in SampEn of IBI | preterm infants measured at 37 to 42 weeks
  Difference in SampEn of IBI in preterm infants measured at 37 to 42 weeks postconceptional age vs. SampEn of IBI in term healthy control infants

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schulzke, Prof. Dr. med, Principal Investigator — University Children's Hospital Basel, UKBB
Locations (1):
- University Children's Hospital Basel UKBB, University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Kaempfen S, Hug M, Sanchez C, Delgado-Eckert E, Schulzke SM. Heart Rate Variability Does Not Predict Recurrence of Apnoea of Prematurity After Ceasing Caffeine Therapy: A Prospective Cohort Study. Acta Paediatr. 2025 Jun;114(6):1371-1378. doi: 10.1111/apa.17579. Epub 2025 Jan 13. PMID 39805735